CLINICAL TRIAL: NCT04104178
Title: A Randomized Placebo-controlled Double-blinded Trial of the Treatment of MRSA Throat Carriage With Either Standard Decolonization Therapy or Standard Decolonization Therapy Combined With Oral Clindamycin
Brief Title: Optimal Treatment of MRSA Throat Carriers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Mona Katrine Alberthe Holm, Coordinating Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MRSATHROAT_2019
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: MRSA; MRSA Colonization
MeSH Terms: interventions — Clindamycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: It's a double blinded placebo study. Only the pharmacy knows the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clindamycin (Active Comparator): 600 mg clindamycin, 3 times daily for 10 days, orally
  Interventions: Drug: Clindamycin
- Placebo (Placebo Comparator): Arm consumes placebo capsules identical to clincamycin capsuls from the other arm,3 times daily for 10 days, orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clindamycin — Investigating whether a significantly higher number of MRSA throat carriers succeed in becoming MRSA free, when using Clindamycin on top of our general recommended topical treatment of Mupirocin nasal ointment + chorhexidin baths
  Other Names: Dalamycin
  Arms: Clindamycin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the optimal way to treat MRSA throat carriers.

DETAILED DESCRIPTION:
The bacterium Staphylococcus aureus frequently colonizes the human skin and mucous membranes. Longitudinal studies usually divide S. aureus carriers into either persistent or intermittent carriers, but because the number of samplings, the follow-up periods and the study populations differ between studies, the designation of carrier state is inconsistent. It has been estimated that around 20 % of a population are persistent carriers, 60 % are intermittent carriers and 20 % are non-carriers. S. aureus is an opportunistic pathogen that can become invasive and cause a large spectrum of infections. S. aureus is frequently the cause of skin and soft tissue infections e.g. wounds, furuncles and abscesses, and can also cause urinary tract infections and pneumonia. If it enters the bloodstream, it can lead to metastatic infections e.g. endocarditis, arthritis, osteomyelitis and meningitis. Furthermore, S. aureus is a common pathogen in surgical site infections and in infections related to foreign bodies, such as catheters and prostheses.

Antibiotic resistance in bacteria is an increasing challenge worldwide and is also seen in S. aureus. The first methicillin resistant Staphylococcus aureus (MRSA) were seen in 1961 just one year after the antibiotic methicillin was introduced. For several decades MRSA was mainly a hospital-associated bacterium, but since the mid 1990's it has become increasingly prevalent in the community where it often affects children and younger adults. MRSA can cause the same types of infections as the methicillin susceptible S. aureus, but often only colonizes the mucosa. When colonization is confirmed, the person is called a carrier of MRSA and there is a risk of both a wide spectrum of infections and spread of MRSA to others. The Danish Health Authority has published a National guideline on how to prevent the spread of MRSA and keep the prevalence of MRSA low in Denmark, especially in the health care setting. The finding of MRSA both in samples from clinical infections and in screening samples for MRSA carriage is notifiable and has to be reported to the Danish Patient Safety Authority and Statens Serum Institut, in order to monitor the number of MRSA positive persons in Denmark, potential outbreaks and risk factors for MRSA acquisition. Furthermore, the guideline recommends that MRSA carriers and their household members undergo a five day topical decolonization treatment consisting of nasal mupirocin ointment 2 % three times daily in the nostrils (mupirocin is an antibiotic usually active against MRSA) and chlorhexidine body wash 4 % once daily. Unfortunately, many patients are still MRSA carriers after completing the treatment and especially throat carriers are difficult to clear.

MRSA carriers have routinely been treated since 2009. Our current guideline recommends adding antibiotics to the standard regimen, clindamycin being our first line choice, on the second or third eradication attempt if the patient is a throat carrier and the isolate is clindamycin susceptible. To our knowledge, the only randomized, controlled trial including clindamycin for treatment of MRSA carriage, is a Swedish study that showed a significant effect of standard treatment plus the antibiotic rifampicin in combination with either clindamycin or sulfamethoxazole/trimethoprim compared to standard treatment alone in long-term MRSA carriers. As most of our patients are healthy individuals without infections, adding systemic antibiotics to the decolonization treatment must be considered thoroughly. There is a risk of side effects in the individual patient and prudent use of antibiotics in the era of a rising incidence of antimicrobial resistance is crucial to avoid selection of further resistance. Our group has recently published a retrospective study describing the MRSA treatment data of 164 patients treated in 2013. The study confirmed that throat carriers had a higher treatment failure rate but adding clindamycin to the first eradication attempt did not significantly increase the success rate. However, as there had been no randomization of patients the scientific evidence is low and the fact that there are no published studies using clindamycin as the only antibiotic for MRSA throat carriers, implies the need for a randomized trial on this subject.

Aim To investigate whether a significantly higher number of MRSA throat carriers become MRSA free when adding the oral antibiotic clindamycin to the standard regimen.

Primary endpoint: MRSA negative swabs at 1 month Secondary endpoint: MRSA negative swabs after 6 months

Methods The study is a randomized double blinded placebo-controlled study, including patients ≥18 years old that have tested MRSA positive in their throat after completing one standard topical decolonization treatment.

Recruitment of study subjects Patients are recruited from the Capital Region via MRSA KnowledgeCenter Hvidovre Hospital or MRSA team Herlev Hospital.

Patients have since their first positive MRSA result an active connection to the MRSA KnowledgeCenter Hvidovre Hospital / MRSA team Herlev Hospital either through the hygiene specialist nurses or doctors. Patients often call for support, guidance and treatment plans, and routine letters are often sent out to patients regarding their treatment, control swap results and more. When the department's nurses or doctors have written or oral contact with a patient that could be a possible candidate for the trial, the possibility of participating in the trial will be mentioned and investigator's contact details will be given.

The patient can contact the investigator by phone or email. After first contact with the investigator, and receiving information about the trial, the patient will have a minimum of 48 hours to decide whether he/she is interested in learning more about the project. Patients that respond positively will be invited to a personal meeting at either Hvidovre Hospital or Herlev Hospital, where oral information about the trial and possible side effects will be given to the patient. The meeting will occur in a private and undisturbed room with the door closed. The patient can bring a friend or relative at the meeting if desired. Patients will be offered 24 hours to provide oral and written informed consent in order to secure sufficient time for reflection on study participation. If a patient needs more time to consider entering the trial, more time will be given. Before signing the informed consent form, the investigator will secure that the patient has read and understood the written study information. Every possible study subject that has a personal meeting with the investigator, will be registered in REDcap, a secure web application for managing online databases.

When oral and written consent has been obtained, the subject will receive a randomized eradication package as described below, as well as a diary to fill out during the study from day 1 to 14, asking about compliance and adverse events.

Patient data Patient data will be pseudo-anonymized as each patient will receive a project number. The investigator will on another file in a locked drawer (investigator site file), as well as on a secured electronic file, only accessible for investigators, have access to the real identification of the patient (the CPR number).

Once included in the trial, one eCRF is created for each patient for collection of trial data. This will include the following data:

Project number, date of birth, age, sex, height, weight, relevant medical history/current medication, sites and dates of MRSA positive samples, prior MRSA decolonization treatments, household composition and household members MRSA carrier state, typing and resistance data of the MRSA strain, body mass index, laboratory and investigational results. For sexually active female subjects in the reproductive age, we also record the use of contraceptives.

The CRFs will be stored in the secure web application for managing online databases 'REDCap' which is designed for non-commercial clinical research. Obtained data will be transferred manually by investigators or appointed research nurses to the CRFs.

The eCRF does not contain information on the specific treatment the patient is randomized to as the randomization is done by the pharmacist.

The treatment The subject will receive a randomized eradication package, consisting of mupirocin nasal ointment 2 %, Chlorhexidine Bodywash 4 % and either placebo capsules 2 capsules three times daily for 10 days or clindamycin 300 mg capsules 2 capsules three times daily for 10 days. Placebo and clindamycin are manufactured to look exactly alike by Glostrup pharmacy, who is also in charge of the randomization/blinding of the packages.

An emergency unblinding procedure will be established to allow investigators the option to withdraw the subject from the trial at any given time, in case of an emergency. This could be if a subject experiences serious adverse events, that could be caused by the active treatment. The pharmacist has created individual sealed and securely closed envelopes for each included subject ID available. The investigator can at any time, 24 hours a day, in case of an emergency unblind a subject, to reveal which treatment has been given. The sponsor will be notified within 24 hours.

Besides the oral treatment, the patient follows the standard treatment guidelines for MRSA decolonization.

After the treatment Thirty to sixty days after end of treatment, the subjects will routinely have MRSA control swabs taken by their GP according to the National MRSA guidelines. Subjects will be reminded about this screening test when entering the trial. If control swabs haven't been received within 6 weeks after completing the treatment, an electronic reminder will be send. The swabs are routine samples that will be handled as regular MRSA control samples in the clinical microbiology laboratory at either Hvidovre hospital or Herlev hospital.

Swab results If the patient is MRSA positive one month after the treatment, no further screening samples will be needed for this project. The patient will leave the trial, and if additional treatment is considered by the doctors responsible for the treatment outside the trial, the randomization will be unblinded in order to plan the most optimal treatment, without revealing the investigator about the investigation medicine given prior to the drop out.

If MRSA negative at one month, no unblinding will take place as no new treatment will be planned. The subject will have new control swabs taken at the GP six to eight months after completing the treatment. If negative swabs at 6-8 months, the patient is declared MRSA free according to the National MRSA Guidelines.

Power calculation Anticipation is 30% better eradication success rate in the group receiving standard treatment plus clindamycin compared to the group treated with standard treatment and placebo. Power calculation shows that 31 patients are needed in each group, power being set at 80 %, and significance level at 0.05 %. It is our goal to include 40 patients in each group, as 9 patients in each group is expected to either drop out or be non-compliant to the treatment.

The number of consumed tablets will be reported in the eCFR, to monitor consumption.

The returned capsules, if any, will be returned to the Glostrup pharmacy, for correct destruction.

The relevance of this trial is high. Hundreds of healthy MRSA carriers have been treated with clindamycin in the last decade without a strong scientific evidence of a better effect than standard treatment. It is very relevant to know, whether adding clindamycin to the treatment of throat carriers is superior to the standard treatment. The outcome of this trial will help us understand the most effective way to clear throat carriers of MRSA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* MRSA carriage in the throat after first topical decolonization treatment (regardless of previous swab results)
* Has completed one standard topical decolonization treatment

Exclusion Criteria:

* Pregnant or lactating woman
* Sexually active women in the reproductive age that do not use approved contraceptives (appendix 4)
* Cannot read or speak Danish (the written participant information is in Danish)
* Skin infection or other active infections
* Activity in skin diseases such as eczema or psoriasis.
* MRSA isolate resistant to clindamycin (defined by inhibition zone size < 22 mm using disk diffusion methodology) or resistant to mupirocin
* Allergy to clindamycin, chlorhexidine or mupirocin
* Taking medications that interact with clindamycin according to the medicine information leaflet.
* MRSA active antibiotic treatment within 7 days before inclusion in the study or during study period
* Followed by specialist due to liver disease
* Severe overweight (BMI > 35) or weight < 50 kg
* Indwelling percutaneous permanent devices such as intravenous catheters or urinary tract catheters
* Daily contact with pigs or minks (decolonization therapy is generally not offered, according to The National Board of Health)
* Nursing home resident or health care worker (they have a more frequent control swab regime)
* Not being capable of completing another treatment successfully
* MRSA positive household members younger than 2 years (MRSA positive children below 2 years of age and their household members are generally not offered decolonization treatment according to The National Board of Health)
* MRSA positive household members, where it is judged that further decolonization attempts are not indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
MRSA negative swabs at 1 month | 30-60 days after treatment
  MRSA negative swabs at 1 month

SECONDARY OUTCOMES:
MRSA negative swabs after 6 months | 6-8 months after treatment
  MRSA negative swabs after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mona KA Holm, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
Availability of study results Results will be published as quickly as possible, in anonymous form, so the subjects cannot be identified. The reporting of the study results will follow the CONSORT 2010 statement.The publications will be in the form of scientific articles, in internationally recognized peer-reviewed journals. Both negative, inconclusive and positive results will be published. Data will be kept 5 years after termination of the trial and will then be destroyed.

REFERENCES:
- [Background] VandenBergh MF, Yzerman EP, van Belkum A, Boelens HA, Sijmons M, Verbrugh HA. Follow-up of Staphylococcus aureus nasal carriage after 8 years: redefining the persistent carrier state. J Clin Microbiol. 1999 Oct;37(10):3133-40. doi: 10.1128/JCM.37.10.3133-3140.1999. PMID 10488166
- [Background] Kluytmans J, van Belkum A, Verbrugh H. Nasal carriage of Staphylococcus aureus: epidemiology, underlying mechanisms, and associated risks. Clin Microbiol Rev. 1997 Jul;10(3):505-20. doi: 10.1128/CMR.10.3.505. PMID 9227864
- [Background] JEVONS MP, COE AW, PARKER MT. Methicillin resistance in staphylococci. Lancet. 1963 Apr 27;1(7287):904-7. doi: 10.1016/s0140-6736(63)91687-8. No abstract available. PMID 13957735
- [Background] Lowy FD. Staphylococcus aureus infections. N Engl J Med. 1998 Aug 20;339(8):520-32. doi: 10.1056/NEJM199808203390806. No abstract available. PMID 9709046
- [Background] Authority DH. Guidance on Preventing the Spread of MRSA. December 13. 2016. p. ISBN online: 978-87-7104-854-4
- [Background] 6.Henius AE, Pedersen K, Jensen LB. Danmap 2017. 2017
- [Background] Bagge K, Benfield T, Westh H, Bartels MD. Eradicating MRSA carriage: the impact of throat carriage and Panton-Valentine leukocidin genes on success rates. Eur J Clin Microbiol Infect Dis. 2019 Apr;38(4):683-688. doi: 10.1007/s10096-019-03474-6. Epub 2019 Jan 25. PMID 30684163